CLINICAL TRIAL: NCT05062720
Title: RT-167: Local Consolidative Therapy in Colorectal Cancer
Brief Title: Local Consolidative Therapy in Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is being closed due to lack of accrual
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 20-1010; RT-167 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2021-09-21; First posted 2021-09-30 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Colorectal Cancer Metastatic
Keywords: oligometastatic; colorectal

STUDY DESIGN:
Intervention Model Description: A total of 105 subjects will be randomized in 2:1 ratio into two cohorts that will receive a combination of LCT along with the systemic therapy or systemic therapy alone.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local consolidative therapy (LCT) + systemic therapy (Experimental): Local Consolidative Therapy (LCT) will be defined as surgical resection or stereotactic body radiotherapy (SBRT) or a combination of both strategies
  Interventions: Radiation: Local consolidative therapy
- Systemic therapy alone (Active Comparator): Appropriate second-line systemic therapy, as defined in the NCCN guidelines will be used during study treatment (https://www.nccn.org/professionals/physician_gls/pdf/colon.pdf). The choice of specific regimen will be left to the discretion of the treating oncologist but cannot include other experimental or investigational treatment. Sample appropriate systemic therapies include FOLFOX or FOLFIRI with a biologic agent such as an anti-angiogenic antibody or anti-EGFR antibody.
  Interventions: Radiation: Local consolidative therapy

INTERVENTIONS:
Radiation: Local consolidative therapy — Local Consolidative Therapy (LCT) will be defined as surgical resection or stereotactic body radiotherapy (SBRT) or a combination of both strategies

SUMMARY:
This is a Phase II randomized multisite trial to study the effect of a combination of local consolidative therapy with systemic therapy in subjects with oligometastatic colorectal cancer who have progressed on the first line of therapy.

DETAILED DESCRIPTION:
This is a Phase II randomized multisite trial to study the effect of a combination of local consolidative therapy with systemic therapy in subjects with oligometastatic colorectal cancer who have progressed on the first line of therapy. The primary objective of this study is progression free survival which is defined as time from randomization until disease progression is documented. Response will be evaluated by scans every 3 months (+/- 7 days). Subjects will continue systemic therapy for 6 months and then at the investigator's discretion, disease progression or unacceptable toxicity. Subjects who are not evaluable for the primary endpoint will be replaced. A total of 105 subjects will be randomized in 2:1 ratio into two cohorts that will receive a combination of LCT along with the systemic therapy or systemic therapy alone.

Arm A: LCT + systemic therapy; 70 subjects will be accrued Arm B: Systemic therapy alone; 35 subjects will be accrued

Systemic therapy will be second line chemotherapy as per NCCN guidelines with the choice of drugs at the treating physician's discretion. Crossover to LCT will be allowed at progression for subjects randomized to Arm B.

The study will be opened at a total of 5 sites with a duration of 26 months of accrual and 10 additional months of follow-up, with a total of 36 months. The study will be conducted in 2 phases with an interim analysis conducted when 29 PFS events have been observed to assess futility/ feasibility of the study.

Subjects will have the option of undergoing tumor biopsy and blood sampling before beginning treatment. A correlative study is proposed using the genomic risk group stratification proposed by Pitroda et al.[9] Collected blood will be analyzed at the conclusion of the trial, with the expectation of comparing levels of circulating tumor DNA between baseline and 3-month time-points between subjects in Arms A and B. As this technology is rapidly evolving, we are not specifying the technology that will be used and will use the most effective assay at the time of trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed metastatic colorectal cancer with 1-3 active metastatic lesions irrespective of location. Previously locally treated (e.g. radiation or interventional radiology-based ablated) metastases that have had a 6-month progression free interval per imaging exams, do not count toward the 1-3 active metastases. Adjacent lymph nodes in the same region constitute one active lesion.
* Subjects must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension in accordance with RECIST criteria v. 1.1 as described in detail in section 12.0.
* All sites of metastatic disease must be amenable to either surgical resection or stereotactic body radiotherapy (SBRT).
* The primary lesion may be either intact or previously resected, but if intact must be resected as part of LCT (primary does not count as one of 1-3 sites of metastatic disease).
* Subjects must have received at least one prior line of systemic therapy with a fluoropyrimidine-based regimen for metastatic disease and be candidates for further systemic chemotherapy. Front-line therapy could have been discontinued for disease progression, unacceptable toxicity, or drug holiday, provided that the therapy was discontinued less than six months from study enrollment.
* Age > 18 years.
* ECOG performance status 0 or 1
* Subjects must have normal organ and marrow function as defined below

  * Absolute neutrophil count > 1,500/mcL
  * Platelets > 100,000/mcL
  * Total bilirubin < 2 mg/dL
  * AST/ALT (SGOT/SGPT) < 5X ULN
  * Creatinine < 1.5X ULN OR
  * Creatinine clearance < 50 ml/min/1.73 m2 for subjects with creatinine levels above institutional normal
* Subjects must possess the ability to understand and willingness to sign a written informed consent and HIPAA consent document.

Exclusion Criteria:

* Subjects must not be experiencing toxicity due to prior therapy that has not resolved to ≤Grade 1 by study registration, with the exception of sensory neuropathy related to previous oxaliplatin exposure, alopecia and fatigue.
* >Grade 2 sensory neuropathy
* Subjects must not be receiving any other investigational agents.
* Subjects must not have known central nervous system (CNS) metastases and/or carcinomatous meningitis, either untreated or treated.
* Subjects must not be unfit to receive combination therapy (>/=2 drugs that could include one biologic agent) as determined by the treating physician.
* Subjects must be able to undergo surgical resection and/or SBRT.
* Subjects must not have 4 or more active metastatic sites.
* Subjects must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Any condition or significant co-morbidity that prevents safe surgery or delivery of SBRT
* Subjects must not be pregnant or breast feeding. Refer to section 4.4 for further detail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 6 months
  To assess the impact of local consolidative therapy (LCT) (surgical resection and/or radiotherapy) on the PFS of subjects with oligometastatic colorectal cancer undergoing second-line systemic therapy. PFS- defined as the duration of time from randomization to date of disease progression or death, whichever occurs first. Individuals who are alive and progression free at last follow-up will be considered censored at the time of last tumor assessment.

SECONDARY OUTCOMES:
Overall suvival (OS) | 6 months
  To assess the impact of local consolidative therapy (LCT) (surgical resection and/or radiotherapy) on the overall survival (OS) of subjects with oligometastatic colorectal cancer undergoing second-line systemic therapy. • OS - defined as the duration of time from randomization to date of death. Individuals who are alive at last follow-up will be considered censored at the time of last contact.
Patient reported outcomes (PROs) | 6 months
  To assess patient reported outcomes (PROs) as measured by the EQ-5D-5L instrument. • PRO - defined as the score on the EQ-5D-5L questionnaire, this will be measured at baseline, and then 2 other times after treatment has begun

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meyer, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No